CLINICAL TRIAL: NCT05622266
Title: Comparative Effectiveness of Pulpotomy and Root Canal Therapy in the Management of Mature Permanent Tooth With Irreversible Pulpits: a Randomized Controlled Non-inferiority Clinical Trial
Brief Title: Effectiveness of Pulpotomy in the Management of Mature Permanent Tooth With Irreversible Pulpits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-334
Record Dates: First submitted 2022-11-13; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-09

CONDITIONS: Irreversible Pulpitis; Mature Teeth
Keywords: pulpotomy; root canal therapy
MeSH Terms: interventions — Pulpotomy; Root Canal Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): The removal of a small portion of the vital coronal pulp as a means of preserving the remaining coronal and radicular pulp tissues.
  Interventions: Procedure: Pulpotomy
- Root Canal Therapy (Active Comparator): The complete removal of the vital dental pulp. Any material or combination of materials placed inside a root canal for the purpose of obturating and sealing the canal space.
  Interventions: Procedure: Root Canal Therapy

INTERVENTIONS:
Procedure: Pulpotomy — The patients who are randomly assigned to the experimental group receive pulpotomy.
  Arms: Pulpotomy
Procedure: Root Canal Therapy — The patients who are randomly assigned to the Active Comparator group receive root canal therapy.
  Arms: Root Canal Therapy

SUMMARY:
This study is to evaluate the effectiveness of pulpotomy in mature permanent tooth with irreversible pulpits, and compare the clinical efficacy of pulpotomy and root canal therapy.

DETAILED DESCRIPTION:
At present, root canal therapy ( RCT ) is still the main treatment for mature teeth diagnosed as irreversible pulpitis, but the teeth after RCT become non-vital, losing the immune defense mechanism and regeneration potential of pulp, which is not conducive to the long-term preservation of teeth. The traditional view is that mature permanent teeth with irreversible pulpitis are not indications for pulpotomy. However, with the deepening of pulp biology research and the availability of new pulp capping materials, the effect of pulpotomy is more predictable. Recent studies have shown that pulpotomy for irreversible pulpitis teeth can achieve good results, however, there is a lack of high-quality randomized controlled clinical studies, and the effect of pulpotomy compared with RCT studies rarely reported. Therefore, this project intends to explore the curative effect of pulpotomy on mature permanent teeth with irreversible pulpitis, and analyze the influence of age, tooth position and other factors on its curative effect, broaden the indications of pulpotomy, and establish the indications and standardized operation process of pulpotomy for mature permanent teeth with irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

Intended to participate with this study, and provide informed assent/consent. Aged 18 and 59 years. At least one mature permanent teeth diagnosed as acute pulpitis or chronic pulpitis, and the teeth was in Nolla stage 9 and above by radiographic examination.

To be prepared to appear for follow-up.

Exclusion Criteria:

Allergic to any medications or materials necessary to complete the procedures. The teeth with severe coronal defect that find to be non-restorable. The teeth with full crown restoration. The teeth with root fracture or vertical root fractures. Patients with periodontitis. Patients who are undergoing orthodontic treatment. Patients with dental dysplasia or other oral genetic disorders. Women who are pregnant or lactating, or women who plan to become pregnant in the subsequent 2 years.

Patients with mental disorders. Patients with a history of systemic diseases that may alter immune function.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of pulpotomy and root canal therapy | From baseline to two years
  The teeth were asymptomatic. Clinical examination showed absence of clinical signs of pain and abscess or sinus tract. Radiographic assessment showed absence of periapical radiolucency.

SECONDARY OUTCOMES:
The pulp vitality in pulpotomy group | From baseline to two years
  The pulpal vitality will be assessed through pulpal response to thermal and electric pulp tests in teeth treated with pulpotomy.
Survival rate of teeth | From baseline to two years
  Survival rate of teeth will be evaluated by function and clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Guo, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No